CLINICAL TRIAL: NCT02924415
Title: Future Internet Social and Technological Alignment Research (FISTAR)
Brief Title: Future Internet Social and Technological Alignment Research
Acronym: FISTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Ana María González-Pinto, Medical Doctor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FISTAR
Record Dates: First submitted 2016-09-27; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele-care support (Experimental): Online psychoeducation treatment using new technologies
  Interventions: Behavioral: Tele-care support
- Control group (Active Comparator): Standard care
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Tele-care support — Psychoeducation treatment based on telemedicine
  Arms: Tele-care support
Other: Control group — Standard care
  Arms: Control group

SUMMARY:
Bipolar disorder patients frequently presents recurring episodes and often experience subsyndromal symptoms, cognitive impairment and difficulties in the functioning with a low quality of life, relapses of disease and recurring hospitalization. Early diagnosis and appropriate intervention may play a role in preventing the neuroprogressive course of bipolar illness. The new technologies represent an opportunity to develop psychological standardized treatments using internet devices that minimizing the limitations of face to face treatments because of its accessibility that allow adjusting to the availability of each user. However, although exist many online psychological programs through web and mobile devices for bipolar disorder, there is not evidence about their efficacy and effectiveness due to the variability in measures and methodology used.

DETAILED DESCRIPTION:
Future Internet Social and Technological Alignment Research (FI-STAR) clinical trial is a randomized simple blind evaluation within an European project. FISTAR is developed to compare this technical solution with treatment as usual. Bipolar disorder patients are to be included and randomly assigned to one of two treatment groups: 1) the experimental group (tele-care support) and the control group. Participants in both groups will be evaluated at baseline (pre-treatment) and at post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of bipolar disorder.
* Being aged between 18-50 years.
* Being in remission (euthymic state).
* Being familiarity with new technologies (computer and /or smartphone).
* Being treatment in the mental health network of the Basque Country (Osakidetza).

Exclusion Criteria:

* Having listening, reading or writing problems.
* Having a diagnosis of mental retardation.
* Unavailability of a smartphone.
* Having manic or depressive symptomatology at the time of inclusion (HAMD> 16 and YOUNG> 8).
* Having suicidal ideation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functioning Assessment Short Test (FAST) | baseline-9 weeks
  To analyze the effectiveness of a psychoeducation treatment based on telemedicine versus usual treatment in relation with better functional outcome of bipolar disorder measured by Functioning Assessment Short Test.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) | baseline-9 weeks
  To analyze the improvement of depressive symptoms of patients measured by Beck Depression Inventory .
State-Trait Anxiety Inventory (STAI) | baseline-9 weeks
  To analyze the improvement of anxiety symptoms of patients measured by State-Trait Anxiety Inventory .
Young Mania Rating Scale (YMRS) | baseline-9 weeks
  To analyze the improvement of manic symptoms of patients measured by Young Mania Rating Scale .
Treatment dropout rate | baseline-9 weeks
  To analyze satisfaction with the treatment received and the contact with the health service by treatment dropout rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ana González-Pinto, MD, Study Chair — ANAMARIA.GONZALEZ-PINTOARRILLAGA@osakidetza.eus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Ortega I, Ugarte A, Ruiz de Azua S, Nunez N, Zubia M, Ponce S, Casla P, Llano JX, Faria A, Gonzalez-Pinto A. Online psycho-education to the treatment of bipolar disorder: protocol of a randomized controlled trial. BMC Psychiatry. 2016 Dec 22;16(1):452. doi: 10.1186/s12888-016-1159-0. PMID 28007034